CLINICAL TRIAL: NCT01624454
Title: Osmotic or Large Volume Lavage for Optimal Bowel Preparation - a Single-blind Randomized Trial
Brief Title: Optimal Bowel Cleansing Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SUS-CRAP
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2012-06

CONDITIONS: Bowel Cleansing for Colonoscopy
Keywords: colonoscopy; bowel cleansing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- large volume (Active Comparator): bowel cleansing with PEG
  Interventions: Other: Laxabon
- Osmotic (Active Comparator)
  Interventions: Other: CitraFleet

INTERVENTIONS:
Other: Laxabon — 4 l PEG solution split dose cleansing
  Arms: large volume
Other: CitraFleet — Small volume osmotic bowelcleansing
  Arms: Osmotic

SUMMARY:
Comparison between large volume and osmotic agent lavage for optimal colonoscopy bowel cleansing, randomizing adult outpatients by invitation letter

DETAILED DESCRIPTION:
This randomized quality assurance trial aims to compare cleansing quality of two different principles of colonoscopy lavage. Large volume PEG solutions are considered safe, but cumbersome and inpalatable, while osmotic solutions are generally more acceptable, however, the risk of electrolyte disturbances or renal decompensation may increase.

The study will focus on patient experience and compliance, as well as cleansing quality, endoscopic findings and other technical parameters of the colonoscopy procedure that may be adversely affected by poor bowel cleansing. Three centers will participate, ensuring a diverse patient population. 800 patients are planned for recruitment, but an interim assessment of statistics of the primary aim parameter (bowel cleansing) will be performed to adjust the number.

ELIGIBILITY:
Inclusion Criteria:

* Pts for out-patient colonoscopy
* age 18-80

Exclusion Criteria:

* Active colitis or suspicion thereof (bloody diarrhea, fever and abdominal pain)
* Suspicion of renal insufficiency or ileus/subileus
* Previous colonic surgery
* Pregnancy
* Inability to adhere to cleansing instructions
* Inability to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Bowel cleansing quality | 1 Day

SECONDARY OUTCOMES:
Colonoscopy findings | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Lars Aabakken, prof of med, Principal Investigator — Prof of medicine
Locations (2):
- Norway (2):
  - OUS Rikshospitalet, dept of med gastro, Oslo, Oslo County
  - Sørlandet sykehus, Kristiansand, VestAgder

REFERENCES:
- [Derived] Leitao K, Grimstad T, Bretthauer M, Holme O, Paulsen V, Karlsen L, Isaksen K, Cvancarova M, Aabakken L. Polyethylene glycol vs sodium picosulfate/magnesium citrate for colonoscopy preparation. Endosc Int Open. 2014 Dec;2(4):E230-4. doi: 10.1055/s-0034-1377520. Epub 2014 Oct 24. PMID 26135098